CLINICAL TRIAL: NCT05391100
Title: Screening of Patients With Rheumatoid Arthritis for Interstitial Lung Disease With Radiographic and Labor Methods
Brief Title: Screening of Patients With Rheumatoid Arthritis for Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Collaborators: Medical Imaging Centre- Semmelweis University, Faculty of Medicine (Unknown); Department of Pulmonology, Semmelweis University Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, dr.Kinga Fritsch, MD, Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Other Study IDs: IV/2683-1/2022/EKU
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
Keywords: rheumatoid arthritis; Interstitial Lung Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum for biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The quantitative and qualitative analysis of RA lung involvement in the Hungarian population

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) accounts for a significant proportion of mortality and morbidity in rheumatoid arthritis (RA). The aim of this prospective longitudinal study is to asess the interstitial lung involvement in Hungarian rheumatoid arthritis patients. Laboratory markers, X-ray based imaging methods, pulmonological functional tests, QOL questionnaire and sleep quality assessement questionnaire are used to estimate the interstitial lung disease. Also smaller cross-sectional studies about the imaging parameters and a national register is planned to be created based on these data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of RA

Exclusion Criteria:

* pregnancy, breastfeeding
* previous diagnosis of ILD, lung cancer, registered lung infection in the last 2 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients with regular follow-ups at Polyclinic of Hospitaller Brothers of St. John of God, Budapest
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ILD | From baseline to at least 5 years
  detection of ILD with imaging methods
pattern of ILD | From baseline to at least 5 years
  to characterize the ILD patterns based on imaging methods

SECONDARY OUTCOMES:
Correlation with biomarkers | From baseline to at least 2 years
  correlation of the imaging results with respiratory function, disease activity and laboratory markers

CONTACTS AND LOCATIONS:
Overall Officials: Judit Majnik, MD PhD, Principal Investigator
Locations (3):
- Hungary (3):
  - Buda Hospital of the Hospitaller Order of Saint John of God, Budapest
  - Medical Imaging Centre, Semmelweis University, Budapest
  - Department of Pulmonology, Semmelweis University Faculty of Medicine, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turesson C. Extra-articular rheumatoid arthritis. Curr Opin Rheumatol. 2013 May;25(3):360-6. doi: 10.1097/BOR.0b013e32835f693f. PMID 23425964
- [Background] Dai Y, Wang W, Yu Y, Hu S. Rheumatoid arthritis-associated interstitial lung disease: an overview of epidemiology, pathogenesis and management. Clin Rheumatol. 2021 Apr;40(4):1211-1220. doi: 10.1007/s10067-020-05320-z. Epub 2020 Aug 13. PMID 32794076
- [Background] Avouac J, Amrouche F, Meune C, Rey G, Kahan A, Allanore Y. Mortality profile of patients with rheumatoid arthritis in France and its change in 10 years. Semin Arthritis Rheum. 2017 Apr;46(5):537-543. doi: 10.1016/j.semarthrit.2016.10.007. Epub 2016 Oct 29. PMID 27908535
- [Background] England BR, Hershberger D. Management issues in rheumatoid arthritis-associated interstitial lung disease. Curr Opin Rheumatol. 2020 May;32(3):255-263. doi: 10.1097/BOR.0000000000000703. PMID 32141954
- [Background] Hodnett PA, Naidich DP. Fibrosing interstitial lung disease. A practical high-resolution computed tomography-based approach to diagnosis and management and a review of the literature. Am J Respir Crit Care Med. 2013 Jul 15;188(2):141-9. doi: 10.1164/rccm.201208-1544CI. PMID 23672718
- [Background] Kim EJ, Collard HR, King TE Jr. Rheumatoid arthritis-associated interstitial lung disease: the relevance of histopathologic and radiographic pattern. Chest. 2009 Nov;136(5):1397-1405. doi: 10.1378/chest.09-0444. PMID 19892679
- [Background] Salvatore M, Henschke CI, Yip R, Jacobi A, Eber C, Padilla M, Knoll A, Yankelevitz D. JOURNAL CLUB: Evidence of Interstitial Lung Disease on Low-Dose Chest CT Images: Prevalence, Patterns, and Progression. AJR Am J Roentgenol. 2016 Mar;206(3):487-94. doi: 10.2214/AJR.15.15537. Epub 2015 Dec 23. PMID 26700157
- [Background] Ley S, Fidler L, Schenk H, Durand M, Marras T, Paul N, Shapera S, Mittoo S. Low dose computed tomography of the lung for detection and grading of interstitial lung disease: A systematic simulation study. Pulmonology. 2021 Jan-Feb;27(1):14-25. doi: 10.1016/j.pulmoe.2020.06.004. Epub 2020 Jun 24. PMID 32591280
- [Background] Hata A, Yanagawa M, Honda O, Miyata T, Tomiyama N. Ultra-low-dose chest computed tomography for interstitial lung disease using model-based iterative reconstruction with or without the lung setting. Medicine (Baltimore). 2019 May;98(22):e15936. doi: 10.1097/MD.0000000000015936. PMID 31145365
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Kauczor HU, Baird AM, Blum TG, Bonomo L, Bostantzoglou C, Burghuber O, Cepicka B, Comanescu A, Couraud S, Devaraj A, Jespersen V, Morozov S, Nardi Agmon I, Peled N, Powell P, Prosch H, Ravara S, Rawlinson J, Revel MP, Silva M, Snoeckx A, van Ginneken B, van Meerbeeck JP, Vardavas C, von Stackelberg O, Gaga M; European Society of Radiology (ESR) and the European Respiratory Society (ERS). ESR/ERS statement paper on lung cancer screening. Eur Respir J. 2020 Feb 12;55(2):1900506. doi: 10.1183/13993003.00506-2019. Print 2020 Feb. PMID 32051182
- [Background] Peelen DM, Zwezerijnen BGJC, Nossent EJ, Meijboom LJ, Hoekstra OS, Van der Laken CJ, Voskuyl AE. The quantitative assessment of interstitial lung disease with positron emission tomography scanning in systemic sclerosis patients. Rheumatology (Oxford). 2020 Jun 1;59(6):1407-1415. doi: 10.1093/rheumatology/kez483. PMID 31642912
- [Background] Nagy A, Nagy T, Kolonics-Farkas AM, Eszes N, Vincze K, Barczi E, Tarnoki AD, Tarnoki DL, Nagy G, Kiss E, Maurovich-Horvat P, Bohacs A, Muller V. Autoimmune Progressive Fibrosing Interstitial Lung Disease: Predictors of Fast Decline. Front Pharmacol. 2021 Dec 22;12:778649. doi: 10.3389/fphar.2021.778649. eCollection 2021. PMID 35002713
- [Background] Barczi E, Nagy T, Starobinski L, Kolonics-Farkas A, Eszes N, Bohacs A, Tarnoki AD, Tarnoki DL, Muller V. Impact of interstitial lung disease and simultaneous lung cancer on therapeutic possibilities and survival. Thorac Cancer. 2020 Jul;11(7):1911-1917. doi: 10.1111/1759-7714.13481. Epub 2020 May 13. PMID 32401433
- [Result] Croia C, Bursi R, Sutera D, Petrelli F, Alunno A, Puxeddu I. One year in review 2019: pathogenesis of rheumatoid arthritis. Clin Exp Rheumatol. 2019 May-Jun;37(3):347-357. Epub 2019 May 10. PMID 31111823
- See also: legislation — https://www.hbcs.hu/uploads/jogszabaly/3129/fajlok/EMMI_szakmai_iranyelv_ILD.pdf
- See also: Research Article — https://akjournals.com/view/journals/650/159/43/article-p1741.xml